CLINICAL TRIAL: NCT03579719
Title: A Single-Center, Non-Randomized, Open-Label, One-Sequence, Two-Period Within-Subject Study to Investigate the Effect of Itraconazole on the Pharmacokinetics of Multiple Doses of Balovaptan in Healthy Volunteers
Brief Title: A Study to Investigate the Effect of Itraconazole on the PK of Multiple Doses of Balovaptan in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: WP40609; 2018-001454-10 (EudraCT Number)
Record Dates: First submitted 2018-06-26; First posted 2018-07-09 (Actual); Results first posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — balovaptan; Itraconazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Balovaptan + Itraconzole (Experimental): Dosing in Period 1 was separated by at least a 7 day washout period before dosing starts in Period 2. Participants received the study drugs in 2 periods over a total of 37 days.
  Interventions: Drug: Balovaptan; Drug: Itraconazole

INTERVENTIONS:
Drug: Balovaptan — In Period 1, balovaptan was administered orally once daily (qd) on Days 1 to 10.
  In Period 2, balovaptan was administered qd on Days 6 to 20.
Drug: Itraconazole — In Period 2, 200 mg itraconzole was administered bid for 4 days and qd on Days 5-20, approximately 12 hours apart. On Days 6-20, 200 mg itraconazole was administered qd.

SUMMARY:
This study was a non-randomized, open-label, one-sequence, two-period within-subject study to investigate the effect of CYP3A inhibition on the PK of balovaptan in healthy male and female volunteers using itraconazole as a CYP3A inhibitor. The study was conducted at 1 site in the Netherlands.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects. Healthy status is defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead ECG, hematology, blood chemistry, urinalysis, and serology.
* Body Mass Index of 18 to 30 kg/m2, inclusive.
* For women of childbearing potential: agreement to use at least 2 acceptable contraceptive methods during the treatment period and for 90 days after the last dose of study drug.
* For men: agreement to use contraceptive measures, and agreement to refrain from donating sperm until 90 days after the last dose of study drug.

Exclusion Criteria:

* Female subjects who are pregnant or lactating.
* Any condition or disease detected during the medical interview/physical examination that would render the subject unsuitable for the study, place the subject at undue risk or interfere with the ability of the subject to complete the study in the opinion of the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2018-11-09 (Actual); Study Completion 2018-11-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Pra International Group B.V, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Derks MGM, Wandel C, Young A, Bolt SK, Meyenberg C. Open-Label Assessment of the Effects of Itraconazole and Rifampicin on Balovaptan Pharmacokinetics in Healthy Volunteers. Adv Ther. 2020 Nov;37(11):4720-4729. doi: 10.1007/s12325-020-01491-y. Epub 2020 Sep 15. PMID 32935287

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 1 site in the Netherlands.
Pre-assignment Details: Participants in this study included healthy volunteers.
Groups:
- Balovaptan + Itraconzole: Dosing in Period 1 was separated by at least a 7 day washout period before dosing started in Period 2. Participants received the study drugs in 2 periods over a total of 37 days.
Period: Overall Study
Arm/Group | Balovaptan + Itraconzole
Started | 15
Completed | 14
Not Completed | 1
Not completed — Protocol deviation, pre-existent disease | 1

BASELINE CHARACTERISTICS:
Arm/Group | Balovaptan + Itraconzole
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) for Balovaptan
Description: Cmax is the observed peak analyte concentration obtained directly from the experimental data without interpolation, expressed in concentration units.
Time Frame: Day 10 of Period 1, Day 10 and Day 15 of Period 2
Population: The Pharmacokinetic (PK) analysis population consisted of all subjects who received at least 1 dose of balovaptan. Subjects were excluded from the PK analysis population if they significantly violated the inclusion or exclusion criteria, deviated significantly from the protocol, or if data were unavailable or incomplete.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Balovaptan + Itraconzole
Number analyzed (Participants) | 14
ng/mL
  Balovaptan Day 10 of Period 1 | 31.5 (25.3)
  Balovaptan + itraconazole Day 10 of Period 2 | 125 (27.7)
  Balovaptan + itraconazole Day 15 of Period 2 | 140 (31.7)

2. Primary Outcome: Maximum Plasma Concentration (Cmax) for M2 Metabolite (as Applicable)
Description: as for outcome 1
Time Frame: Day 10 of Period 1, Day 10 and Day 15 of Period 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Balovaptan + Itraconzole
Number analyzed (Participants) | 14
ng/mL
  Balovaptan Day 10 of Period 1 | 11.0 (26.5)
  Balovaptan + itraconazole Day 10 of Period 2 | 6.34 (45.3)
  Balovaptan + itraconazole Day 15 of Period 2 | 7.60 (44.9)

3. Primary Outcome: Maximum Plasma Concentration (Cmax) for M3 Metabolite
Description: as for outcome 1
Time Frame: Day 10 of Period 1, Day 10 and Day 15 of Period 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Balovaptan + Itraconzole
Number analyzed (Participants) | 14
ng/mL
  Balovaptan Day 10 of Period 1 | 19.9 (16.5)
  Balovaptan + itraconazole Day 10 of Period 2 | 21.3 (20.0)
  Balovaptan + itraconazole Day 15 of Period 2 | 28.6 (19.7)

4. Primary Outcome: Area Under the Concentration Vs Time Curve Over the Dosing Interval (AUC0-tau) for Balovaptan
Time Frame: Day 10 of Period 1, Day 10 and Day 15 of Period 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | Balovaptan + Itraconzole
Number analyzed (Participants) | 14
ng.h/mL
  Balovaptan Day 10 of Period 1 | 464 (29.7)
  Balovaptan + itraconazole Day 10 of Period 2 | 2304 (31.8)
  Balovaptan + itraconazole Day 15 of Period 2 | 2587 (35.1)

5. Primary Outcome: Area Under the Concentration Vs Time Curve Over the Dosing Interval (AUC0-tau) for M2 Metabolite (as Applicable)
Time Frame: Day 10 of Period 1, Day 10 and Day 15 of Period 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | Balovaptan + Itraconzole
Number analyzed (Participants) | 14
ng.h/mL
  Balovaptan Day 10 of Period 1 | 230 (26.9)
  Balovaptan + itraconazole Day 10 of Period 2 | 129 (46.9)
  Balovaptan + itraconazole Day 15 of Period 2 | 156 (48.5)

6. Primary Outcome: Area Under the Concentration Vs Time Curve Over the Dosing Interval (AUC0-tau) for M3 Metabolite
Time Frame: Day 10 of Period 1, Day 10 and Day 15 of Period 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | Balovaptan + Itraconzole
Number analyzed (Participants) | 14
ng.h/mL
  Balovaptan Day 10 of Period 1 | 402 (17.8)
  Balovaptan + itraconazole Day 10 of Period 2 | 449 (21.3)
  Balovaptan + itraconazole Day 15 of Period 2 | 570 (20.9)

7. Secondary Outcome: Trough Plasma Concentration (Ctrough) for Balovaptan
Time Frame: Day 10 of Period 1; Day 10 and Day 15 of Period 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Balovaptan + Itraconzole
Number analyzed (Participants) | 14
ng/mL
  Balovaptan Day 10 of Period 1 | 13.3 (4.7)
  Balovaptan + itraconazole Day 10 of Period 2 | 91.9 (26.6)
  Balovaptan + itraconazole Day 15 of Period 2 | 102 (36.0)

8. Secondary Outcome: Trough Plasma Concentration (Ctrough) for M2 Metabolite (as Applicable)
Time Frame: Day 10 of Period 1; Day 10 and Day 15 of Period 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Balovaptan + Itraconzole
Number analyzed (Participants) | 14
ng/mL
  Balovaptan Day 10 of Period 1 | 9.93 (2.62)
  Balovaptan + itraconazole Day 10 of Period 2 | 5.82 (2.99)
  Balovaptan + itraconazole Day 15 of Period 2 | 6.88 (3.05)

9. Secondary Outcome: Trough Plasma Concentration (Ctrough) for M3 Metabolite
Time Frame: Day 10 of Period 1; Day 10 and Day 15 of Period 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Balovaptan + Itraconzole
Number analyzed (Participants) | 14
ng/mL
  Balovaptan Day 10 of Period 1 | 15.1 (2.5)
  Balovaptan + itraconazole Day 10 of Period 2 | 18.9 (4.7)
  Balovaptan + itraconazole Day 15 of Period 2 | 23.9 (6.1)

10. Secondary Outcome: Time to Steady State for Balovaptan
Time Frame: Days 1, 3, 5, 8, 9, 10 in Period 1 and Days 1, 3, 5, 8, 9, 10, 13, 14, 15 in Period 2
Population: as for outcome 1
Measure: Number; unit: Day
Arm/Group | Balovaptan + Itraconzole
Number analyzed (Participants) | 14
Day
  Balovaptan | 4
  Balovaptan + itraconazole | 13

11. Secondary Outcome: Percentage of Participants With Adverse Events
Time Frame: Up to 21 days postdose
Population: The safety analysis population consisted of subjects who received at least one dose of balovaptan.
Measure: Number; unit: Percentage
Arm/Group | Balovaptan + Itraconzole
Number analyzed (Participants) | 15
Percentage | 73

12. Primary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) for Balovaptan
Time Frame: Day 10 of Period 1; Day 10 and Day 15 of Period 2
Population: as for outcome 1
Measure: Median (Full Range); unit: Hour(s)
Arm/Group | Balovaptan + Itraconzole
Number analyzed (Participants) | 14
Hour(s)
  Balovaptan Day 10 of Period 1 | 3.00 [1.00 to 6.00]
  Balovaptan + itraconazole Day 10 of Period 2 | 4.00 [2.00 to 10.00]
  Balovaptan + itraconazole Day 15 of Period 2 | 4.00 [2.00 to 24.00]

13. Primary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) for M2 Metabolite (as Applicable)
Time Frame: Day 10 of Period 1; Day 10 and Day 15 of Period 2
Population: as for outcome 1
Measure: Median (Full Range); unit: Hour(s)
Arm/Group | Balovaptan + Itraconzole
Number analyzed (Participants) | 14
Hour(s)
  Balovaptan Day 10 of Period 1 | 5.00 [0.00 to 12.00]
  Balovaptan + itraconazole Day 10 of Period 2 | 6.00 [0.00 to 24.00]
  Balovaptan + itraconazole Day 15 of Period 2 | 6.00 [0.00 to 24.00]

14. Primary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) for M3 Metabolite
Time Frame: Day 10 of Period 1; Day 10 and Day 15 of Period 2
Population: as for outcome 1
Measure: Median (Full Range); unit: Hour(s)
Arm/Group | Balovaptan + Itraconzole
Number analyzed (Participants) | 14
Hour(s)
  Balovaptan Day 10 of Period 1 | 4.00 [1.00 to 24.00]
  Balovaptan + itraconazole Day 10 of Period 2 | 9.00 [2.00 to 24.00]
  Balovaptan + itraconazole Day 15 of Period 2 | 3.50 [1.00 to 8.00]

ADVERSE EVENTS:
Time Frame: From the first study drug to the data cutoff date: 9 Nov 2018 (up to 21 days postdose)
Arm/Group | Balovaptan + Itraconzole
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 11/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Balovaptan + Itraconzole (N=15)
Headache (Nervous system disorders) | 3
Head discomfort (Nervous system disorders) | 2
Presyncope (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Medical device site pruritus (General disorders) | 1
Asthenia (General disorders) | 2
Catheter site pain (General disorders) | 2
Catheter site haematoma (General disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Anal pruritus (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Insomnia (Psychiatric disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-05-18): https://cdn.clinicaltrials.gov/large-docs/19/NCT03579719/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-20): https://cdn.clinicaltrials.gov/large-docs/19/NCT03579719/SAP_001.pdf